CLINICAL TRIAL: NCT00475553
Title: The Frequency and Management of Breakthrough Bleeding During Extended Therapy With the Transvaginal Contraceptive Ring
Brief Title: Management of Breakthrough Bleeding During Extended Therapy Use With NuvaRing®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scott and White Hospital & Clinic (Other)
Collaborators: Organon (Industry)
Responsible Party: Dr. Patricia Sulak, Scott and White Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 50403
Record Dates: First submitted 2007-05-16; First posted 2007-05-21 (Estimated); Last update posted 2009-12-18 (Estimated); Status verified 2009-12

CONDITIONS: Breakthrough Bleeding; Breakthrough Spotting
Keywords: spotting; PMS; nuvaring; birth control; pelvic pain; headache; mood swings; continuous use
MeSH Terms: conditions — Metrorrhagia; Pelvic Pain; Headache | interventions — etonogestrel; Ethinyl Estradiol; NuvaRing; Contraceptive Devices, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 2 (Other): Subject will use the nuvaring and if they developed breakthrough bleeding or spotting for more than 5 days on the 6th day the ring would be removed and would leave it out for 3 full days and reinsert the same ring the next day. All subjects would be filling out a daily diary or calendar which would rate their blood flow, pelvic pain, headaches, moods, how many pain pills were taken and how many pads, liners or tampons would be used.
  Interventions: Other: remove ring if bleeding or spotting occurs more than 5 days
- Group 1 (Other): Subject is using the nuvaring continuously and it would be changed out monthly. If she develops breakthrough bleeding or spotting she does not remove the ring until it is her time to change it. All subjects would be filling out a daily diary or calendar which would rate their blood flow, pelvic pain, headaches, moods, how many pain pills were taken and how many pads, liners or tampons would be used.
  Interventions: Other: If bleeding does not remove ring

INTERVENTIONS:
Other: remove ring if bleeding or spotting occurs more than 5 days — Both groups of women will be using the nuvaring continuously, ie if the ring is placed on 3rd of January, on the 3rd of February the ring would be removed and a new one inserted. On the 3rd of March the same thing would happen and so forth. Group 2 if bleeding or spotting occurs for more than 5 days then on the 6th day the ring is removed and will keep it out for three more days and reinsert the same ring on the 4th day.
  Other Names: etonogestrel/ethinyl estradiol
  Arms: Group 2
Other: If bleeding does not remove ring — Subject is using the nuvaring continuously. For example she puts the ring in on 3rd of January then the 3rd of February is when that ring is removed and another one is inserted. The 3rd of March the same thing occurs.
  Other Names: nuvaring; etonogestrel/ethinyl estradiol; vaginal ring
  Arms: Group 1

SUMMARY:
The purpose of this research study is to evaluate the best way to manage breakthrough spotting and bleeding during an extended use regimen of NuvaRing®. Ease of use and acceptability of a flexible regimen of NuvaRing® will also be evaluated. A comparison of cyclic mood symptoms, pelvic pain, and headaches will be made between a standard 21/7 regimen and an extended regimen.

DETAILED DESCRIPTION:
Hormonal contraception is undergoing a change away from a 21/7 day regimen where a woman utilizes a combination estrogen and progestin therapy for 21 days followed by 7 days of a hormone-free interval (HFI). It is well documented that women may experience a higher incidence of mood changes, headaches and cramping that begin prior to and during this 7 day HFI. By reducing the HFI and extending the active combination contraceptive therapy, it is hoped that women will experience greater satisfaction with their contraceptive regimen and will experience fewer negative side effects associated with a HFI.

The most common reason for discontinuation of an extended contraception regimen is irregular bleeding. The purpose of this research study is to evaluate the best way to manage this breakthrough spotting and bleeding. Ease of use and acceptability of a flexible regimen of NuvaRing will also be evaluated. A comparison of cyclic mood symptoms, pelvic pain, and headaches will be made between a standard 21/7 regimen and an extended regimen.

The contraceptive ring used in this study contains both an estrogen (ethinyl estradiol) and a progestin (etonogestrel). These are synthetic (man-made) hormones. The amount of ethinyl estrogen released into the bloodstream each day is 120mcg and the amount of etonogestrel is 150mcg. The NuvaRing®, by Organon, is FDA approved for contraception, but is not approved for use in an extended regimen. Therefore its use in this study is considered investigational.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years of age
* Currently utilizing combination estrogen/progestin contraception for a period of at least 2 months or 1 month if previously using a progestin only pill.

Exclusion Criteria:

* Body Mass Index (BMI) of 38 or greater
* Anyone who should not be using hormonal contraception due to contraindications
* Anyone who smokes > 10 cigarettes per day or if 35 years old or older smokes any cigarettes
* Anyone who is taking antiretroviral therapy (due to many drug interactions)
* Women using other estrogen-containing products or herbal products that contain phytoestrogens
* Known or suspected pregnancy, or desiring pregnancy in the next year

Additionally, NuvaRing® should not be used in women who currently have the following conditions:

* Thrombophlebitis
* A past history of deep vein thrombophlebitis or thromboembolic disorders
* Cerebral vascular or coronary artery disease (current or history)
* Valvular heart disease with thrombogenic complications
* Severe hypertension
* Diabetes with vascular involvement
* Headaches with focal neurological symptoms
* Major surgery in patients with prolonged immobilization
* Known or suspected carcinoma of the breast or personal history of breast cancer
* Carcinoma of the endometrium or other known or suspected estrogen dependent neoplasia
* Undiagnosed abnormal genital bleeding
* Cholestatic jaundice of pregnancy or jaundice with prior hormonal contraceptive use
* Hepatic tumors (benign or malignant) or active live disease
* Hypersensitivity to any components of NuvaRing®

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2006-05; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
a comparison of days and extent per day of bleeding and spotting within subjects for continuous use pattern of nuvaring. | 6 months

SECONDARY OUTCOMES:
a comparison of choice to switch patterns or stick with randomized pattern for second phase of study (2nd 6 month interval). | 6 months
comparisons of all symptoms (pelvic pain, headaches, moodiness, and pain medication use) both within subjects during different treatment intervals and between subject groups. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Sulak, MD, Principal Investigator — Scott and White Hospital & Clinic
Locations (1):
- Scott & White Hospital and Clinic, Temple, Texas, United States